CLINICAL TRIAL: NCT01143012
Title: Group Eczema Education Visits:Impact on Patient and Family Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Susan Tofte, Principal Investigator, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Group eczema education visits
Record Dates: First submitted 2010-06-09; First posted 2010-06-14 (Estimated); Last update posted 2019-07-11 (Actual); Status verified 2019-07

CONDITIONS: Eczema
Keywords: Group eczema education
MeSH Terms: conditions — Eczema | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group eczema education session (Active Comparator): One group will attend a group eczema education session. All subjects will answer quality of life questions two times.
  Interventions: Other: Group eczema education session
- Control group (Active Comparator): The other group will not attend the group eczema education session. Both groups will be asked quality of life questions two times.
  Interventions: Other: Control group

INTERVENTIONS:
Other: Group eczema education session — Subjects in the intervention group will participate in a group education visit to discuss topics such as subjects' general understanding and knowledge of eczema and its treatment.
  Arms: Group eczema education session
Other: Control group — The control group will not attend the group eczema education session.
  Arms: Control group

SUMMARY:
The objective of this study is to determine whether group educational visits improve the quality of life of patients referred to the Dermatology Clinic. Secondary outcomes will be to determine whether group educational visits influences other key elements of patient care such as topical steroid usage, disease exacerbations, emergency visits, and phone calls to the office. Lastly, the investigators hope to evaluate which aspects of the educational visit were found to be the most helpful to families caring for children with atopic dermatitis (AD). Patients will be new atopic dermatitis referrals to OHSU dermatology and pediatric dermatology clinics. All consecutive patients with such appointments during a three month time period will be screened for participation in the study. Parents will be recruited via telephone. In the intervention group, parents will be invited to participate in a group education visit prior to their first appointment with a dermatologist. All parents in the study will fill out questionnaires. The children involved in the study will be assigned an eczema severity score during their routine visits, but this will be incorporated into the regular clinic assessment. The Childhood Atopic Dermatitis Impact Scale (CADIS) assesses the quality of life in households with children who have atopic dermatitis. The Eczema Area and Severity Index (EASI) measures the extent and severity of the patient's atopic dermatitis. The change in CADIS scores will be analyzed to determine if there is a more significant improvement in quality of life for the group in which parents receive the group eczema education visit.

ELIGIBILITY:
Inclusion Criteria:

* Children ages 2 months though 6 years.
* Participants must carry a diagnosis of atopic dermatitis according to the Hanifin and Rajka criteria.
* New patients or consultations at an OHSU clinic.
* English-speaking families will be included in this study

Exclusion Criteria:

* Subjects who have been on systemic therapies for treatment of their atopic dermatitis (prednisone or cyclosporine)

Ages: 2 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2010-05; Primary Completion 2011-08 (Actual); Study Completion 2014-04-13 (Actual)

PRIMARY OUTCOMES:
The difference between the two groups in CADIS score | 4 weeks
  The primary outcome will be the difference between the two groups in CADIS score as measured at four weeks. CADIS is a validated outcome of pediatric quality of life in AD.

SECONDARY OUTCOMES:
Assess extent of skin disease. | Between 4 weeks and 4 months of the first visit.
  EASI (Eczema Area and Severity Index) scores will be performed to assess extent of skin disease at an interval between 4 weeks and 4 months of the first visit.
Assess average monthly number of follow-up phone calls. | Between 4 weeks and 4 months of the first visit.
  A chart review will be done to assess average monthly number of follow-up phone calls.
Assess average monthly number of urgent and emergency visits. | Between 4 weeks and 4 months of the first visit.
  A chart review will be done to assess average monthly number of urgent and emergency visits.

CONTACTS AND LOCATIONS:
Overall Officials: Susan J. Tofte, FNP-C, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States